CLINICAL TRIAL: NCT05310721
Title: Efficacy and Feasibility of Time-restricted Eating on Cardiometabolic Health in Adults With Overweight/Obesity: The EXTREME Study
Brief Title: Efficacy and Feasibility of Time-restricted Eating on Cardiometabolic Health in Adults With Overweight/Obesity
Acronym: EXTREME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Universidad Pública de Navarra (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXTREME
Record Dates: First submitted 2022-01-17; First posted 2022-04-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Time Restricted Feeding; Obesity, Abdominal; Cardiometabolic Syndrome
MeSH Terms: conditions — Intermittent Fasting; Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early time-restricted eating (Experimental): Participants will eat ad libitum within an 8-hour early eating window. The first meal will be before 10 am (last meal before 18h). No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Interventions: Behavioral: Early time-restricted eating
- Late time-restricted eating (Experimental): Participants will eat ad libitum within an 8-hour late eating window. The first meal will be at 13h or later (last meal not before 21h). No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Interventions: Behavioral: Late time-restricted eating
- Self-selected time-restricted eating (Experimental): Participants will self-selecte an 8-hour eating window to eat ad libitum. No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Interventions: Behavioral: Self-selected time-restricted eating
- Usual-care group (No Intervention): Participants will receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion

INTERVENTIONS:
Behavioral: Early time-restricted eating — Participants will eat ad libitum within an 8-hour early eating window starting not later than 10am. No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Arms: Early time-restricted eating
Behavioral: Late time-restricted eating — Participants will eat ad libitum within an 8-hour late eating window starting not earlier than 1pm. No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Arms: Late time-restricted eating
Behavioral: Self-selected time-restricted eating — Participants will self-selected an 8-hour eating window to eat ad libitum. No calorie-containing food or beverage intake will be allowed outside the 8-hour eating window. Participants will also receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion
  Arms: Self-selected time-restricted eating

SUMMARY:
In Spain, obesity epidemic is one of the leading contributors of chronic disease and disability. Obesity is associated with higher morbidity and all-cause mortality risk especially when fat is stored in the abdominal area (i.e., increased visceral adipose tissue, VAT). Although current approaches such as energy restriction may be effective at reducing body fat and improving cardiometabolic health, their long-term adherences are limited. Time-restricted eating (TRE; e.g., 8 hours eating: 16 hours fasting on a daily basis) is a recently emerged intermittent fasting approach with promising cardiovascular benefits. Results from pioneering pilot studies in humans are promising and suggest that simply reducing the eating time window from ≥12 to ≤8-10 hours/day improves cardiometabolic health. However, currently, there is no consensus regarding whether the TRE eating window should be aligned to the early or middle to late part of the day. The EXTREME study will investigate the efficacy and feasibility of three different 8 hours TRE schedules (i.e., early, late and self-selected) over 12 weeks on VAT (main outcome) and cardiometabolic risk factors (secondary outcomes) in adults with overweight/obesity and abdominal obesity. The final goal of the EXTREME study is to demonstrate the health benefits of a novel and pragmatic intervention for the treatment of obesity and related cardiometabolic risk factors; an approach readily adaptable to real-world practice settings, easy for clinicians to deliver, and intuitive for patients to implement and maintain in their lives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-60 years.
* Body mass index ≥25.0 and <40 kg/m2
* Weight stability (within 3% of screening weight) for >3 months prior to study entry.
* Sedentary lifestyle (<150 min/week of moderate-vigorous intensity exercise) for >3 months prior to study entry.
* Habitual eating window ≥12 hours.
* At least one of the following metabolic impairments:

  * High-density lipoprotein (HDL) cholesterol concentration <50 mg/dL for females and <40 mg/dL for males.
  * Low-density lipoprotein (LDL) cholesterol levels >100 mg/dL (or on medication to treat elevated LDL cholesterol levels).
  * Serum triglycerides concentration ≥150 mg/dL or on medication to treat elevated triglycerides.
  * Systolic blood pressure >130 mm Hg and/or diastolic blood pressure >85 mm Hg or already being treated with anti-hypertension medications.
  * Impaired glucose tolerance is defined as at least one of the following:

    * Fasting plasma glucose (PG) >100 mg/dL and <125 mg/dL.
    * Hemoglobin A1c between ≥5.7% and <6.5%.
    * Insulin resistance as measured by the Homeostatic Model Assessment of Insulin Resistance (HOMA2-IR) >1.8.

Exclusion Criteria:

* History of a major adverse cardiovascular event, clinically significant kidney, endocrine, or neurological disease, bariatric surgery, HIV/AIDS, known inflammatory and/or rheumatologic disease, cancer, or other medical condition in which fasting or exercise is contraindicated.
* Type 1 or Type 2 diabetes.
* Major psychiatric disorders, eating disorders, sleep disorders, or alcohol abuse.

Regular use of medication or compounds that may affect study outcomes (e.g., antidiabetic, steroids, beta-blockers, antibiotics, prebiotics, probiotics and symbiotics).

* Participating in a weight loss or a weight-management program.
* Pregnancy and lactation or planned pregnancy (within the study period).
* Caregiver for a dependent requiring frequent nocturnal care/sleep interruptions. Shift workers with variable hours (e.g., nocturnal). Frequent travel over time zones during the study period.
* Fear of needles and claustrophobia to magnetic resonance imaging (MRI).
* Being unable to understand and to accept the instructions or the study objectives and protocol.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Change in visceral adipose tissue | Change from baseline to 12 weeks
  Visceral adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Change in Hepatic fat content | Change from baseline to 12 weeks
  Hepatic fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in Pancreatic fat content | Change from baseline to 12 weeks
  Pancreatic fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in Intramuscular fat content | Change from baseline to 12 weeks
  Intramuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in Hepatic elasticity | Change from baseline to 12 weeks
  Hepatic elasticity will be assessed by US elastography
Change in Pancreatic elasticity | Change from baseline to 12 weeks
  Pancreatic elasticity will be assessed by US elastography
Change in Fasting glucose metabolism | Change from baseline to 12 weeks
  Fasting blood samples will be used to analyse different biomarkers of glucose metabolism
Change in Fasting lipid metabolism | Change from baseline to 12 weeks
  Fasting blood samples will be used to analyse different biomarkers of lipid metabolism (e.g., triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol)
Change in Inflammatory profile | Change from baseline to 12 weeks
  Fasting blood samples will be used to analyse inflammatory profile (e.g., C-reactive protein and interleukin 6)
Change in Hepatic profile | Change from baseline to 12 weeks
  Fasting blood samples will be used to analyse hepatic profile (e.g., alkaline phosphatase, bilirubin, alanine transaminase and gamma-glutamyl transferase)
Change in Kidney profile | Change from baseline to 12 weeks
  Fasting blood samples will be used to analyse kidney profile (e.g., creatinine and creatine kinase)
Change in Glycemia (Continuous Glucose Monitoring) | Change from baseline to 12 weeks
  Glycemia will be assessed by Continuous Glucose Monitoring during 2 weeks
Change in Body weight | Change from baseline to 12 weeks
  Body weight will be measured by a digital scale
Change in Body composition (Fat mass and fat free mass) | Change from baseline to 12 weeks
  Body composition will be assessed by Dual-energy X-ray Absorptiometry (DXA)
Change in Anthropometric measures | Change from baseline to 12 weeks
  Neck, hip and waist circumferences will be assessed by standard procedures
Change in Blood pressure | Change from baseline to 12 weeks
  Systolic and Diastolic blood pressure will be assessed by standard procedures
Change in energy intake | Change from baseline to 12 weeks
  Energy intake (kcal/day) will be assessed by 24h recalls
Change in macronutrients intake | Change from baseline to 12 weeks
  Macronutrients intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in dietary habits | Change from baseline to 12 weeks
  Dietary habits will be assessed by food frequency questionnaires
Change in Food craving | Change from baseline to 12 weeks
  Food craving will be assessed by the Food Craving Inventory (FCI)
Change in Appetitive traits | Change from baseline to 12 weeks
  Appetitive traits will be assessed by the Adult Eating Behavior Questionnaire (AEBQ)
Change in Subjective sleep quality | Change from baseline to 12 weeks
  Subjective sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI)
Change in Objectively sleep quality | Change from baseline to 12 weeks
  Objectively sleep quality will be assessed by accelerometry
Change in Chronotype | Change from baseline to 12 weeks
  Chronotype will be assessed by the Munich Chronotype Questionnaire (MCTQ)
Change in Morning-Evening type | Change from baseline to 12 weeks
  Morning-Evening type will be assessed by the Morningness-Eveningness Questionnaire Self-Assessment Version.
Change Subjective physical activity levels | Change from baseline to 12 weeks
  Subjective physical activity levels will be assessed by the International Physical Activity Questionnaire short form
Change Objectively physical activity levels | Change from baseline to 12 weeks
  Objectively physical activity levels will be assessed by accelerometry
Change in Depression aspects | Change from baseline to 12 weeks
  Depression aspects will be assessed by the Beck Depression Inventory Fast Screen (BDI-FS)
Change in Stress aspects | Change from baseline to 12 weeks
  Stress aspects will be assessed by the Perceived Stress Scale (PSS)
Change in Anxiety aspects | Change from baseline to 12 weeks
  Anxiety aspects will be assessed by the State-Trait Anxiety Inventory (STAI)
Change in General health | Change from baseline to 12 weeks
  General health will be assessed by the EuroQol 5 dimensions 5 levels (EQ-5D-5L)
Change in Quality of life | Change from baseline to 12 weeks
  Quality of life will be assessed by the Rand Short Form 36 (SF-36)
Change in Gut microbiota composition | Change from baseline to 12 weeks
  DNA sequencing to determine gut microbiota composition (e.g., phylum and genera)
Change in Gut microbiota diversity | Change from baseline to 12 weeks
  DNA sequencing to determine gut microbiota diversity (e.g., beta and alpha)
Feasibility of recruitment | 12 weeks
  Feasibility of recruitment (i.e., percent of response rate).
Feasibility of the intervention | 12 weeks
  Retention during the intervention (i.e., percent of attrition).
Adherence to the intervention | Every day during the intervention, up to 90 days
  Adherence will be assessed by eating records
Genetic variants in Clock genes | Baseline
  Genetic variantes in clock genes will be determined by Illumina sytem

OTHER OUTCOMES:
Epigenetic changes in clock genes | Change from baseline to 12 weeks
  Changes in selected CpG in clock genes will be determined by Illumina system

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan R. Ruiz, PhD, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - Universidad Pública de Navarra, Pamplona, Navarre
  - University of Granada, Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clavero-Jimeno A, Dote-Montero M, Migueles JH, Camacho-Cardenosa A, Medrano M, Alfaro-Magallanes VM, Oses M, Carneiro-Barrera A, de Cabo R, Munoz-Torres M, Labayen I, Ruiz JR. Time-Restricted Eating and Sleep, Mood, and Quality of Life in Adults With Overweight or Obesity: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2517268. doi: 10.1001/jamanetworkopen.2025.17268. PMID 40560588
- [Derived] Dote-Montero M, Clavero-Jimeno A, Merchan-Ramirez E, Oses M, Echarte J, Camacho-Cardenosa A, Concepcion M, Amaro-Gahete FJ, Alcantara JMA, Lopez-Vazquez A, Cupeiro R, Migueles JH, De-la-O A, Garcia Perez PV, Contreras-Bolivar V, Munoz-Garach A, Zugasti A, Petrina E, Alvarez de Eulate N, Goni E, Armendariz-Brugos C, Gonzalez Cejudo MT, Martin-Rodriguez JL, Idoate F, Cabeza R, Carneiro-Barrera A, de Cabo R, Munoz-Torres M, Labayen I, Ruiz JR. Effects of early, late and self-selected time-restricted eating on visceral adipose tissue and cardiometabolic health in participants with overweight or obesity: a randomized controlled trial. Nat Med. 2025 Feb;31(2):524-533. doi: 10.1038/s41591-024-03375-y. Epub 2025 Jan 7. PMID 39775037